CLINICAL TRIAL: NCT02379845
Title: A Multicenter Randomized, Open-Label Phase II/III Study, To Compare The Efficacy Of NBTXR3, Implanted As Intratumor Injection And Activated By Radiotherapy, Versus Radiotherapy Alone In Patients With Locally Advanced Soft Tissue Sarcoma Of The Extremity And Trunk Wall
Brief Title: NBTXR3 Crystalline Nanoparticles and Radiation Therapy in Treating Randomized Patients in Two Arms With Soft Tissue Sarcoma of the Extremity and Trunk Wall
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Nanobiotix (Industry)
Collaborators: PharmaEngine (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NBTXR3-301
Record Dates: First submitted 2015-02-19; First posted 2015-03-05 (Estimated); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Adult Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental): NBTXR3 + Radiotherapy
  Interventions: Device: NBTXR3; Device: Radiation therapy
- Arm B (Active Comparator): Radiotherapy alone
  Interventions: Device: Radiation therapy

INTERVENTIONS:
Device: NBTXR3 — One intratumor implantation by injection
  Other Names: PEP503
  Arms: Arm A
Device: Radiation therapy — 5 weeks/50 Gy (5 x 2 Gy by week)

SUMMARY:
RATIONALE: Radiation therapy given before surgery of soft tissue sarcoma decreases the size of the tumor mass and the presence of malignant cells in its peripheral region. NBTXR3 and radiation therapy may kill more cancer cells and increase the tumor shrinkage rendering surgery more feasible or easier and achieve better local control of the tumor.

PURPOSE: This phase II/III is a prospective randomized, multi-center, open-label and active controlled two arms study in patients with locally advanced soft tissue sarcoma (STS) of the extremity and trunk wall. Patients will be randomized to receive either NBTXR3 as intratumor injection, activated by external beam radiation therapy or external beam radiation therapy alone, as preoperative treatment. Once the radiotherapy treatment is completed, tumor surgery will be performed in all patients.

DETAILED DESCRIPTION:
Patients who will be allocated in arm A, will receive a single intratumor injection of NBTXR3 and will receive external beam radiotherapy starting 24hrs after the injection up to completion of 5 weeks, 5 days a week of treatment (50Gy, 2Gy/fraction). Then, all patients will undergo surgical resection of the tumor 5 weeks later and will be followed for wound healing and toxicity assessment. A visit of end of treatment will take place approximately 3-4 weeks after surgery. Patients will be followed for evaluation of their disease status and adverse event until the end of study.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years and older
* Locally Advanced Soft Tissue Sarcoma of the Extremity and Trunk Wall
* All grades
* Candidate to radiotherapy + surgery (ESMO guideline 2014) i.e. tumor must not have involvement of bone and / or vessel and or nerve :

  * Primary tumor or,
  * Relapsed tumor, localized out of previously irradiated area
* WHO performance score 0 to 2
* Adequate function of bone marrow
* Adequate renal function
* Adequate hepatic function
* Adequate pulmonary function
* All female patients of childbearing potential must have a negative serum/urinary pregnancy test

Exclusion Criteria:

* Absence of written Informed Consent duly signed and dated
* Patients with the following histological type: embryonal or alveolar rhabdomyosarcoma, Ewing's sarcoma, osteosarcoma or chondrosarcoma, Kaposi's sarcoma, primitive neuroectodermal tumor, angiosarcoma, aggressive fibromatosis or dermatofibrosarcoma protuberans
* Soft Tissue Sarcoma of the Trunk Wall localized in the abdominal region i.e. the region defined cranially by the xiphoid process of the sternum and the costal margins, and caudally by the line joining the anterior superior iliac spines, both limited by the perpendicular lines crossing both nipples
* Patient with a calculated tumor baseline volume > 3000 mL
* Metastatic disease (CT-scan / MRI verification) with life expectancy shorter than 6 months
* Previous radiation therapy in relapse site of soft tissue sarcoma (no radiation re-challenge is permitted)
* Concurrent treatment with any other anticancer therapy, including chemotherapy, immunotherapy, targeted therapy, gene therapy, or patients planning to receive these treatments during the study
* Absence of histologically or cytologically proven cancer at the first diagnosis
* Previous neoadjuvant chemotherapy treatment given as an upfront of the current treatment line
* Hemolytic anemia
* Autoimmune disease
* Complete initial work up earlier than 4 weeks prior to patient registration
* Patients unable to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures
* Patients participating in another clinical investigation at the time of signature of the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2015-03-03 (Actual); Primary Completion 2018-05-22 (Actual); Study Completion 2020-09-20 (Actual)

PRIMARY OUTCOMES:
Pathological Complete Response Rate (pCRR) | 36 months
  To compare antitumor activity in terms of Pathological complete response rate (pCRR) of intratumor injection of NBTXR3 activated by external beam radiation therapy (EBRT), versus EBRT alone

SECONDARY OUTCOMES:
Incidence of early and late TEAE, post-TEAE, SAE and laboratory abnormalities (NCI CTCAE V4.0) | 36 months
Objective Response Rate (ORR) by Imaging (MRI) according to RECIST 1.1 | 36 months
Tumor volume changes (theoretical tumor volume estimated as: Length x Width x Depth | 36 months
Resection Margins (R0, R1, R2) | 36 months
Hyalinization, fibrosis, necrosis and tumor infarction percentage | 36 months
Limb amputation rate | 36 months

OTHER OUTCOMES:
Local and distant recurrence rate | 12 months and 24 months

CONTACTS AND LOCATIONS:
Locations (42):
- Australia (2):
  - Capital Region Cancer Service, Canberra Hospital, Canberra
  - Chris O'Brien Lifehouse, Sydney
- Belgium (2):
  - Jules Bordet Institute, Brussels
  - Ghent University Hospital, Ghent
- France (9):
  - Centre Rene Gauducheau, Nantes, Saint Herblain
  - Institut Bergonie, Bordeaux
  - Centre Leon Berard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Centre Regional de Lutte Contre Le Cancer Paul Lamarque, Montpellier
  - Centre Antoine Lacassagne, Nice
  - Institut Curie, Paris
  - Institut Claudius Regaud - Oncopole, Toulouse
  - Institut Gustave Roussy, Villejuif
- Germany (2):
  - Klinikum Mannheim, Mannheim
  - Klinikum Nürnberg, Nuremberg
- Princes of Wales Hospital, Shatin, Hong Kong
- Hungary (3):
  - Medical Centre, Hungarian Defence Forces, Budapest
  - National Institute of Oncology, Budapest
  - University Pècs, Pécs
- Italy (3):
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Institute of Oncology Veneto IOV, Padua
  - Instituto Nazionale Tumori Regina Elena, Rome
- Oslo University Hospital, Oslo, Norway
- Philippines (4):
  - Perpetual Succour Hospital Cebu, Cebu City
  - University of Santo Thomas, Manila
  - The Medical City, Pasig
  - St. Luke's Medical Center, Quezon City
- Cancer Center Institute, Warsaw, Poland
- Romania (6):
  - Institutul Oncologic Bucuresti, Bucharest
  - Spitalului Universitar de Urgenta Militar Central, Bucharest
  - Amethyst-Cluj, Floreşti
  - County Hospital 'Dr Gavril Curteanu', Oradea
  - County Hospital, Targu Mures, Târgu Mureş
  - Municipal Emergency Hospital, Timișoara
- South Africa (4):
  - Iatros International, Bloemfontein
  - The Oncology Centre, Durban
  - Gvi Outeniqua Oncology Unit, George
  - Wilgers Oncology Centre, Pretoria
- Spain (4):
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Hospital Clinico Universitario San Carlos, Madrid
  - START MADRID, Hospital Fundacion Jimenez Diaz, Madrid
  - START MADRID, Hospital Universitario Madrid Norte Sanchinarro, Madrid

REFERENCES:
- [Derived] Bonvalot S, Rutkowski PL, Thariat J, Carrere S, Ducassou A, Sunyach MP, Agoston P, Hong A, Mervoyer A, Rastrelli M, Moreno V, Li RK, Tiangco B, Herraez AC, Gronchi A, Mangel L, Sy-Ortin T, Hohenberger P, de Baere T, Le Cesne A, Helfre S, Saada-Bouzid E, Borkowska A, Anghel R, Co A, Gebhart M, Kantor G, Montero A, Loong HH, Verges R, Lapeire L, Dema S, Kacso G, Austen L, Moureau-Zabotto L, Servois V, Wardelmann E, Terrier P, Lazar AJ, Bovee JVMG, Le Pechoux C, Papai Z. NBTXR3, a first-in-class radioenhancer hafnium oxide nanoparticle, plus radiotherapy versus radiotherapy alone in patients with locally advanced soft-tissue sarcoma (Act.In.Sarc): a multicentre, phase 2-3, randomised, controlled trial. Lancet Oncol. 2019 Aug;20(8):1148-1159. doi: 10.1016/S1470-2045(19)30326-2. Epub 2019 Jul 8. PMID 31296491